CLINICAL TRIAL: NCT01419379
Title: Epidemiologic Review and Prospective Observation of COPD and Health in Korea
Brief Title: This is a Multicenter, Prospective and Retrospective and Descriptive Epidemiology Study in Patients With Chronic Obstructive Pulmonary Disease (COPD) in Korea
Acronym: EPOCH
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-401-KR; U1111-1142-0154 (Registry Identifier: WHO)
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: COPD
Keywords: COPD exacerbation rate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study is designed as a multicenter, prospective and retrospective and descriptive epidemiology study.

This study is planned to evaluate 2 years of exacerbation in COPD patients and to investigate correlation of COPD disease progress and its exacerbation.

This study is designed with 6 months of subject enrollments, 12 months of retrospective study, and 12 months of prospective study. Hence, each patient will be participating in the study for 12 months, while the actual data collections from the patients will take a total of 24 months.

The statistical analysis of this study will be done twice, at the completion of 1 year retrospective data collection and at the completion of next 1 year follow-up.

The 1st statistical analysis of retrospective study includes exacerbation rate, duration of hospitalization for exacerbation and lung function test for the past 1 year from the enrollment and comorbidities, COPD assessment (CAT) and COPD medication at the enrollment will be analyzed.

The 2nd statistical analysis of prospective 1-year follow-up includes changes in exacerbation rates, comparison of lung function test results, comorbidities, COPD assessments (CAT) and COPD medications of retrospective and prospective studies for the 2 years as well as mortality rate.

ELIGIBILITY:
Inclusion Criteria:

1. Over 40 years old
2. Patient with at least 1 year of medical history of COPD as defined by GOLD criteria
3. Patient with having past 1 year medical record at the investigational site
4. Patient who signed Informed Consent Form

Exclusion Criteria:

1. Patients who are currently involved in any other interventional studies or possible to be involved for the next 1 year
2. Patients currently diagnosed with cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Probability Sample
Enrollment: 1118 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To investigate exacerbation rate in patients suffering from COPD | 24 months
  A total of 2 years of data will be evaluated based on annual evaluations:
  * 1 year-before the enrollment (past 1 year) and
  * 1 year-after the enrollment (1 year from the enrollment)

SECONDARY OUTCOMES:
To investigate comorbidities of COPD | At screening and after 12 months
To determine airflow obstruction through lung function test | 24 months
  Lung function test data will be collected at the time of enrollment, 1 year before the enrollment (if available) and 1 year after the enrollment.
  For lung function data, the closest ones to the evaluation date among those obtained from ±3 months will be used.
  Items to be collected are pre/post bronchodilator FEV1, FVC, FEV1/FVC.
To assess COPD (through CAT) | At screening and after 12 months
  Patients will complete CAT (COPD Assessment Test) questionnaire.
To know the current use of medications for COPD treatment | At screening and after 12 months
  Medications for COPD treatment at the time of enrollment will be investigated.
To investigate mortality of COPD patients for 1 year period | 12 months

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Nycomed Investigational Site, Busan
  - Nycomed Investigational Site, Chungcheongnam-do
  - Nycomed Investigational Site, Daegu
  - Nycomed Investigational Site, Daejeon
  - Nycomed Investigational Site, Gangwon-do
  - Nycomed Investigational Site, Gwangju
  - Nycomed Investigational Site, Gyeongbuk
  - Nycomed Investigational Site, Gyeonggi-do
  - Nycomed Investigational Site, Gyeongsangnam-do
  - Nycomed Investigational Site, Incheon
  - Nycomed Investigational Site, Jeollanam-do
  - Nycomed Investigational Site, Jeonbuk
  - Nycomed Investigational Site, Seoul
  - Nycomed Investigational Site, Ulsan